CLINICAL TRIAL: NCT03306966
Title: Assessing the Safety and Performance of the Single Use Endoscopic Linear Cutter Stapler and Reloads (Frankenman) in Colectomy: a Monocentric Post-market Observational Study
Brief Title: Assessing the Safety and Performance of the Endoscopic Linear Cutter Stapler and Reloads (Frankenman) in Colectomy
Status: Withdrawn | Type: Observational
Why Stopped: Design modification
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-02
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-03

CONDITIONS: Colon Cancer
Keywords: Ascending colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colon cancer patients: Patients with colon cancer (ascending colon) eligible for laparoscopic or open segmental colectomy.
  Interventions: Device: Endoscopic Linear Cutter Stapler and Reloads (Frankenman)

INTERVENTIONS:
Device: Endoscopic Linear Cutter Stapler and Reloads (Frankenman) — The Single Use Endoscopic Linear Cutter Stapler and Reloads from Frankenman received CE-mark in April 2013. It is used to staple and simultaneously divide tissue from the central line.

SUMMARY:
The purpose of this observational study is to evaluate the safety and performance of the Single Use Endoscopic Linear Cutter Stapler and Reloads from Frankenman used in (hemi)colectomy to remove tumors and create anastomoses in patients with cancer in the ascending colon. The goal of the study will be achieved by assessing the device performance and reporting of peri- and postoperative complications in a prospectively maintained database.

ELIGIBILITY:
Inclusion Criteria:

* Age at study entry is at least 18 years.
* Patient must sign and date the informed consent form prior to the index-procedure.
* Patient has a tumor in the ascending colon.

Exclusion Criteria:

* Patient is pregnant.
* Patient has inflammatory bowel disease (ulcerative colitis, Crohn's disease).
* Patient has symptomatic diverticulitis.
* Patient has bowel trauma.
* Patient has peritoneal carcinomatosis.
* Patient is known to be, or suspected of being unable to comply with the study protocol or proposed follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer (ascending colon) eligible for laparoscopic or open segmental colectomy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events related to the index-procedure. | 3 to 4 weeks follow-up
  Determination of peri- and postoperative anastomotic leaks and intra-intestinal/intra-abdominal bleeding.
Number of patients with adverse events related to the index-procedure. | 3 months follow-up
  Determination of peri- and postoperative anastomotic leaks and intra-intestinal/intra-abdominal bleeding.
Number of patients with adverse events related to the index-procedure. | 6 months follow-up
  Determination of peri- and postoperative anastomotic leaks and intra-intestinal/intra-abdominal bleeding.

SECONDARY OUTCOMES:
Number of adverse device effects. | 3 to 4 weeks follow-up
  Determination of the sharpness of the blade and occurrence of disruption of the staple line.
Number of adverse device effects. | 3 months follow-up
  Determination of the sharpness of the blade and occurrence of disruption of the staple line.
Number of adverse device effects. | 6 months follow-up
  Determination of the sharpness of the blade and occurrence of disruption of the staple line.
Number of patients with peri- and early/late postoperative complications related to the open and laparoscopic colectomy. | 3 to 4 weeks follow-up
Number of patients with peri- and early/late postoperative complications related to the open and laparoscopic colectomy. | 3 months follow-up
Number of patients with peri- and early/late postoperative complications related to the open and laparoscopic colectomy. | 6 months follow-up
Number of patients with colectomy related re-interventions. | 3 to 4 weeks follow-up
Number of patients with colectomy related re-interventions. | 3 months follow-up
Number of patients with colectomy related re-interventions. | 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Van Der Speeten, Dr, Principal Investigator — ZOL, Genk